CLINICAL TRIAL: NCT02472015
Title: Dementia in Long Term Care Facilities: Telemedicine for the Management of Neuropsychiatric Symptoms.
Acronym: DETECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 13 7031 08
Record Dates: First submitted 2015-06-01; First posted 2015-06-15 (Estimated); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Dementia
Keywords: neuropsychiatric symptoms; dementia; telemedicine; long-term care facilities
MeSH Terms: conditions — Dementia | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- normal care (No Intervention): patients who will have normal care
- telemedicine (Experimental): patients who will have telemedicine
  Interventions: Procedure: telemedicine

INTERVENTIONS:
Procedure: telemedicine — psycho-behavioural care by telemedicine
  Arms: telemedicine

SUMMARY:
Telemedicine may facilitate adequate treatment of Neuropsychiatric symptoms (NPS) by identifying underlying causes and tailoring a treatment plan (pharmacological or non-pharmacologic treatments including provision of staff education and support, training in problem solving, and targeted therapy directed at the underlying causes for specific behaviors).

DETAILED DESCRIPTION:
During a 6-months period, patients will be included in both arms, whenever they present a disruptive NPS that requires a specialist consultation based on the long-term care facility (LTCF) staff judgment. In the intervention group, a telemedicine (TM) consultation between the LTCF staff (medical and nurse staff) and the Memory Center from the University Hospital, will occur at inclusion (T0). Then, a second TM consultation will occur at 1 month (T1). In the control group management of NPS will be done as usual care. In both groups, patients' parameters such as non-programmed hospitalizations and/or consultations due to disruptive NPS, psychotropic drugs use, and health costs, will be evaluated at inclusion, 1 month and at 2 months. Acceptability of the TM among the LTCF staff will be assessed during the study in the intervention group.

The two university hospitals are composed of a group of institutions for elderly people located near Toulouse and Limoges.

ELIGIBILITY:
Inclusion Criteria:

* patient aged 65 or more, with a dementia diagnosed by a specialist or the general practitioner;
* patient presenting with a disruptive NPS as defined in French Haute Autorité de Santé (HAS) recommendations (2009), that requires a specialist consultation based on the LTCF staff judgment;
* informed and written consent by the patient or the legal representative or the reliable person when appropriate;
* general practitioner agreement.

Exclusion Criteria:

* patient's life expectancy less than 6 months;
* Non agreement of study participation of patients or legal representative or the reliable person when appropriate.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 143 (Actual)
Dates: Start 2015-06; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Acceptability of the TM among the LTCF staff | 6 months
  Acceptability of the telemedicine (TM) among the LTCF staff which will be assessed in the intervention group by quantitative indicators (proportion of the solicitation of the TM solution among patients with disruptive NPS, the delay to obtain a TM consultation and the number of the staff participants at each TM consultation) and qualitative indicators (staff global satisfaction will be evaluated by focus groups and interviewing).

SECONDARY OUTCOMES:
Rate of non-programmed hospitalizations and/or consultation due to disruptive NPS | 6 months
  Calculation of the rate of non-programmed hospitalizations and/or consultation due to disruptive NPS in both groups
The psychotropic drugs used | 6 months
  Description of psychotropic drugs used in both groups
describe the health costs | 6 months
  Description of the health costs in both groups
describe the estimation of the cluster effect ("design effect") | 6 months
  Estimation of the cluster effect ("design effect") in both groups

CONTACTS AND LOCATIONS:
Overall Officials: Maria Soto, MD, Principal Investigator — University Hospital, Toulouse
Locations (2):
- France (2):
  - UHLimoges, Limoges
  - UHToulouse, Toulouse

REFERENCES:
- [Background] Piau A, Nourhashemi F, De Mauleon A, Tchalla A, Vautier C, Vellas B, Duboue M, Costa N, Rumeau P, Lepage B, Soto Martin M. Telemedicine for the management of neuropsychiatric symptoms in long-term care facilities: the DETECT study, methods of a cluster randomised controlled trial to assess feasibility. BMJ Open. 2018 Jun 12;8(6):e020982. doi: 10.1136/bmjopen-2017-020982. PMID 29895651
- [Result] Piau A, Vautier C, De Mauleon A, Tchalla A, Rumeau P, Nourhashemi F, Soto-Martin M. Health workers perception on telemedicine in management of neuropsychiatric symptoms in long-term care facilities: Two years follow-up. Geriatr Nurs. 2020 Nov-Dec;41(6):1000-1005. doi: 10.1016/j.gerinurse.2020.07.009. Epub 2020 Aug 6. PMID 32771311